CLINICAL TRIAL: NCT02277158
Title: A Phase I Study of Concurrent Radiotherapy and Tegafur, Gimeracil and Oteracil Potassium Capsule(S-1) as Adjuvant Treatment for Stage II/III Operable Rectal Cancer.
Brief Title: Phase I Study of CCRT as Adjuvant Treatment for Stage II/III Operable Rectal Cancer.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhen-zhou Yang, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP03182014
Record Dates: First submitted 2014-10-22; First posted 2014-10-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; S-1; Chemoradiotherapy; Phase I
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemoradiotherapy (Experimental): There are four dose levels and one arm only. Level 1: S-1, 50 mg/m2, Day 1-14, 22-35; RT Total dose 50.4Gy/28fractions/6 weeks Level 2: S-1, 65 mg/m2, Day 1-14, 22-35; RT Total dose 50.4Gy/28fractions/6 weeks Level 3: S-1, 80 mg/m2, Day 1-14, 22-35; RT Total dose 50.4Gy/28fractions/6 weeks Level 4: S-1, 90 mg/m2, Day 1-14, 22-35; RT Total dose 50.4Gy/28fractions/6 weeks
  Interventions: Drug: Chemoradiotherapy

INTERVENTIONS:
Drug: Chemoradiotherapy — S-1 CCRT

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and safety of S-1 plus radiotherapy for patients with rectal cancer

DETAILED DESCRIPTION:
This stage I study is designed to evaluate the appropriate dose of S-1 plus radiotherapy for patients with R0 resection of rectal cancer for stage II-III patients(AJCC 7th). To evaluate safety, data on adverse events will be collected from the time of enrollment until withdrawn of complete whole study.

ELIGIBILITY:
Inclusion Criteria:

* R0 resection of histologically proved stage II/III rectal cancer;
* 18-75 years old;
* No previous radiotherapy or chemotherapy for rectal cancer;
* Performance status of ECOG 0,1;
* Adequate organ function defined as below:

  i. WBC ≥ 4,000/mm^3 ii. ANC ≥ 1,500/mm^3 iii. Hemoglobin ≥ 10g/dL iv. Platelet ≥ 100,000/m^3 v. Total bilirubin ≤ 1.5ULN vi. AST/ALT ≤ 1.5ULN vii. Serum creatinine ≤ 1.5ULN or creatinine clearance rate ≥ 60ml/min、Urea nitrogen ≤ 1.5ULN viii. Protein in urine dipstick test<1+; if the test result >1+ ,total protein in urea must <500mg within 24 hours
* Able to receive oral administration
* Informed consent

Exclusion Criteria:

* Hypersensitive to S-1 or its excipients
* Pulmonary fibrosis or interstitial pneumonitis found within 28 days prior to registration
* Significant co-morbid medical conditions, including, but not limited to, heart failure, renal failure, hepatic failure, hemorrhagic peptic ulcer, mechanical or paralytic ileus, or poorly controlled diabetes
* Received any investigational drug or anti-cancer agent
* Pregnant or lactating female or pregnancy test positive
* Severe mental disorder
* Judged ineligible by physicians for participation in the study due to safety concern.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 6weeks (42 days)

SECONDARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | 6weeks (42 days)
Quality of Life | 6weeks (42 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenzhou-Yang, Chongqing, Chongqing Municipality, China